CLINICAL TRIAL: NCT05324969
Title: The Feasibility and Preliminary Efficacy of the Mindful-Healthy Family Intervention With Rural Families
Acronym: MHFproject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Tsui-Sui A Kao, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006180
Record Dates: First submitted 2022-03-14; First posted 2022-04-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: intervention group will receive 9 intervention sessions (via zoom or phone call) every other week and 3 texts/week to motivate lifestyle changes. Three times of rescheduling is allowed. Attention control group will receive 9 biweekly emails about other health related topics.
Who Masked: Participant
Masking Description: No marking intended given low budget and fewer research assistants available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MM-based MI group (Experimental): Intervention group parents will receive 9 intervention sessions every other week by trained staff via 9 online sessions via Zoom or phone calls. Each intervention session will last 30-40 minutes. Intervention group parents will receive 3 text messages per week. No in-person contacts will be conducted without MSU department permission. All assessments will be delivered remotely with guided phone calls or zoom conference. The assessment of dyads' BMI, %BF, and WC will be obtained remotely from the parents using the scale and measuring tape delivered to their home.
  Interventions: Behavioral: MM-based MI
- Control group (Other): Control group parents will receive a total of 9 emailed packets of educational materials (without information related to the mindfulness-based motivational interviewing [MM-based-MI]). The pre and post assessments will be collected the same way as the participants at intervention group.
  Interventions: Other: healthy education

INTERVENTIONS:
Behavioral: MM-based MI — 9 remote mindful-based MI sessions will be delivered to promote participating parents' mindful eating, mindful movements, and mindful family interactions. Parents will be encouraged to act as changing agents for their families.
  Arms: MM-based MI group
Other: healthy education — 9 health education emails will be sent to participating parents in the control group
  Arms: Control group

SUMMARY:
This two-group RCT, the Mindful-Healthy Family project, will test the feasibility and preliminary efficacy of a mindfulness-based Motivational Interviewing (MM-based-MI) intervention with rural families within Michigan. This two-group RCT will enroll 34-60 families from Michigan rural or suburban communities with one OW/O parent-figure adult (BMI ≥25) who has at least one child (ages 3-6) at home. The targeted parents will serve as the change agent. The outcome assessments include BMI and optional hair cortisol as well as parent's collective family efficacy, perceived stress, depression score, 24 hours dietary recall (ASA24; healthy eating index [HEI]), mindful eating score, Physical Activity (IPAQ-short) at both baseline and post-intervention. These intervention group families will receive 9 online sessions (30 min/session) delivered via Zoom or phone calls every other week by trained research staff. BMI will be obtained directly from the participating parents using the scale delivered to their homes. Attention control arm families will have same assessment and will receive a total of 9 mailed packets of educational materials. This work will advance the science by explicating how MM and MI work synergistically.

DETAILED DESCRIPTION:
The RCT aims to enroll 34-60 families from Michigan rural or suburban communities. Because the investigators are targeting overweight or obese parents (BMI greater than 25 but less than 45),the investigators anticipate excluding some ineligible families. The investigators plan to use the rolling admission strategy to obtain eligible families. With our inclusion/exclusion criteria, the investigators estimate the needs to approach approximately 80-300 parents. To begin, the investigators will start the eligibility screening and recruitment procedure with local community recruiters from willing clinics, rural communities as well as online advertisements. If the investigators do not have a sufficient sample by the end of two months, the investigators will proceed to recruit families from rural communities to suburban communities via Craigslist advertisements and other online platforms. The investigators will use our previous experience with the rural communities to determine strategies needed to proceed with our recruitment effort.

In fall 2022, The investigators will hire 2-3 part-time staffs from the Tribal communities to assist us with recruitment efforts with American Indian families. The investigators would also use snowball any eligible families identified by our enrolled families. This local part-time staff will distribute recruitment flyer to adjunct American Indian communities. Potential participants can complete eligibility screening either by a self-administered online survey (Qualtrics) or by direct interactions with research staff (either in-person or telephone calls).

Intervention Procedure:

The outcome assessments (BMI and optional hair cortisol assessments) as well as surveys (ASA24 and Qualtrics) will be collected remotely. The RA will call the participating families and guide assessment step by step using the measurement tool sent to their homes. Once enrolled, participating families will be randomized into two groups (1.5 to 1 ratio): intervention and control group.

Intervention group parents will also receive nine intervention sessions every other week by trained research staff. The investigators will deliver the intervention via 9 online sessions delivered via Zoom or phone calls. Each intervention session will last about 30-40 minutes. Interventional group parents will receive 3 text messages (or emails, per preference) per week to improve their motivation to lead a mindful and healthy lifestyle (eating, physical activity, and positive family interactions). No in-person contacts will be conducted without MSU department permission. The assessment of dyads' BMI will be obtained directly and remotely from the participating parents using the scale and measuring tape delivered to their homes. Hair cortisol assessment is optional for the participants. If willing, the participants will receive a hair sample collection video as well as written instruction. A step-by step assistance (via phone call or zoom) will be available for participants. Control group parents will receive a total of 9 emailed packets of educational materials (without information related to the mindfulness-based motivational interviewing [MM-based-MI]). Assessment procedure remains the same for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-11 years old and one of his/her parent whose BMI >25 but less than 45.
* Both parent and child are required to enroll together
* Parent and child are willing to do height and weight assessment (using the scale and wall growth chart mailed to home) and some surveys (parents only) remotely

Exclusion Criteria:

* excluding participants who are pregnant at baseline.
* exclude mentally and/or physically disabled person.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Parents' Healthy Eating Index (HEI) converted from ASA24 | changes from baseline to post intervention about 4-6 months after baseline
  Automated Self-Administered 24-Hour Dietary Assessment (ASA24 2020) tool at NIH

SECONDARY OUTCOMES:
Optional Hair Cortisol (dyads) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  Hair Cortisol (optional and only when in-person assessment is allowed)
Parents' Physical Activity | change from baseline to post intervention, about 4-6 months after baseline assessment.
  self-reported Physical Activity (PA) using the International Physical Activity Questionnaire (IPAQ). The minimal score is 0 and the maximal score is 4,000 MET-minutes. A higher score represents a higher intensity of physical activity.
health literacy (parent only) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  using the Newest Vital Sign to assess parents' healthy literacy
Kids' food screeners (parents reporting kids' eating pattern) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  Block Kids food screeners to assess kids' eating patterns
Child's Physical Activity | change from baseline to post intervention, about 4-6 months after baseline assessment.
  This is one item survey assessing the children's Physical Activity in the past 7 day. The minimal score is 0 day and the maximal score is 7 days/week. A higher score represents a higher number of days in the past week that the child spent at least 60 minutes a day.
Self-efficacy for Exercise (parents) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  This is 9-item self-reported self-efficacy measure. A 10-item perceived stress scale (0-4 Likert scale). The minimal score is 0 and the maximal score is 40. A higher score represents a higher level of perceived stress.
Collective family efficacy (parents) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  This is a 20-item collective family efficacy scale (1-7-point Likert scale). The minimal score is 20, and the maximal score is 140. A higher score represents a higher level of collective family efficacy.
Centre for Epidemiological Studies Depression Scale (CES-D10) | change from baseline to post intervention, about 4-6 months after baseline assessment.
  Centre for Epidemiological Studies Depression Scale (CES-D 10) will be used to assess parents' depression symptoms. This is a 10-item depression symptom scale. The minimal score is 0, and the maximal score is 30. A higher score represents greater depressive symptoms.
Parents' perceived stress | change from baseline to post intervention, about 4-6 months after baseline assessment.
  This is a 10-item perceived stress scale will be used to assess parents' perceived stress level. The minimal score is 0, and the maximal score is 60. A higher score represents greater depressive symptoms.
Parent's family function | change from baseline parent's family function scores about 4-6 months after baseline assessment
  This is a 5-item family function scale assessing family member's Adaptability, Partnership, Growth, Affection, and Resolve. The minimal score is 0, and the maximal score is 10. A higher score represents a greater satisfaction of family functioning in above five domains.
Mindful eating questionnaire | change from baseline parent's mindful eating scores at 4 -6 months after baseline assessment.
  This is a 28-item 1-4-point scale assessing parent's mindful eating attitudes in four domains (awareness, distraction, disinhibition, emotional, external). The subsumed score will be divided by the item number allocated in each domain. The minimal score is 1, and the maximal score is 4. A higher score represents a higher level of mindful eating in each domain.
Parent BMI | change from baseline BMI at 4 -6 months after baseline assessment.
  Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Tsui-Sui A Kao, PhD, Principal Investigator — MSU College of Nursing
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
in our approved IRB application, there is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Kao TA, Ling J, Alanazi M, Bara N, Barnes Najor J. Feasibility and preliminary effects of the mindful healthy family project among rural families. Health Psychol Behav Med. 2024 Dec 26;13(1):2446368. doi: 10.1080/21642850.2024.2446368. eCollection 2025. PMID 39777051